CLINICAL TRIAL: NCT03249207
Title: Does Interleukin-1 Receptor Antagonist Improve Outcome Following Aneurysmal Subarachnoid Haemorrhage (aSAH)? A Phase III Trial
Brief Title: SC IL-1Ra in SAH - Phase III Trial (SCIL)
Acronym: SCIL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Clinical Trials Unit, Manchester (Other); Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R121178
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL-1Ra twice daily (Active Comparator)
  Interventions: Drug: IL-1Ra
- Placebo twice daily (Placebo Comparator)
  Interventions: Drug: IL-1Ra Placebo

INTERVENTIONS:
Drug: IL-1Ra — Doses to be administered subcutaneously (SC) twice daily (12 hourly) starting within 72 hours of ictus (onset of symptoms) for a maximum of 21 days from ictus (or sooner if discharged from neurosurgical centre).
  Arms: IL-1Ra twice daily
Drug: IL-1Ra Placebo — Doses to be administered subcutaneously (SC) twice daily (12 hourly) starting within 72 hours of ictus (onset of symptoms) for a maximum of 21 days from ictus (or sooner if discharged from neurosurgical centre).
  Arms: Placebo twice daily

SUMMARY:
This phase III trial will establish whether IL-1Ra, with sub-cutaneous (SC) administration twice daily for up to 21 days post aneurysmal subarachnoid haemorrhage (aSAH), improves clinical outcome as measured by ordinal shift in mRS at 6 months.

Patients with SAH transferred to a neurosurgical centre will be identified and approached for study participation. Following consent, patients will be randomised to receive either IL-1Ra or placebo for a maximum of 21 days from onset of symptoms. Patients who are found to be non-aneurysmal following randomisation will be withdrawn from the study treatment. Blood samples for plasma IL-6 will be obtained prior to randomisation and at day 3-5 post randomisation for IL-6 & IL-1 measurement. Safety will be measured at 30 days post randomisation and outcome assessed at 6 months post randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CT positive spontaneous SAH admitted to a participating neurosurgical centre where written informed consent can be obtained and study drug can be administered within 72 hours of ictus.
2. No concomitant health problems that, in the opinion of the PI or designee, would interfere with participation, administration of study drug or assessment of outcomes including safety.
3. Willing and able to give informed consent or consent available from a patient representative for trial inclusion including agreement in principle to receive study drug and undergo all study assessments.
4. Male or female aged 18 years or above.

Exclusion Criteria:

1. Unconfirmed or uncertain diagnosis of spontaneous SAH.
2. Known active tuberculosis or active hepatitis.
3. Known active malignancy.
4. Known Still's Disease
5. Neutropenia (ANC <1.5 x 109/L ).
6. Abnormal renal function (creatinine clearance or estimated Glomerular Filtration Rate (eGFR) < 30 ml/minute) documented in the last 3 months prior to this SAH.
7. Live vaccinations within the last 10 days of this SAH.
8. Previous or concurrent treatment with IL-1Ra known at the time of trial entry or previous participation in this trial.
9. Current treatment with TNF antagonists.
10. Known to have participated in a clinical trial of an investigational agent or device in the 30 days prior to ictus.
11. Known to have participated in a clinical trial of an investigational agent or device within 5 half-lives (of the previous agent or device) prior to ictus.
12. Known to be pregnant or breast feeding or inability to reliably confirm that the patient is not pregnant
13. Clinically significant serious concurrent medical condition, pre morbid illnesses, or concurrent serious infection, at the PI's (or designee's) discretion, which could affect the safety or tolerability of the intervention.
14. Known allergy to IL-1Ra or any of the excipients listed in the drug SmPC
15. Known allergy to other products that are produced by DNA technology using the micro-organism E. coli (e.g. E.coli derived protein).
16. Current treatment with IL-6 or IL-1 inhibitors or drugs affecting the IL-1 axis.
17. History of DRESS syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Ordinal shift in modified Rankin Score (mRS) | 6 months post randomisation

SECONDARY OUTCOMES:
Measurement of mood using HADS | 6 months post randomisation
Measurement of fatigue using Fatigue score | 6 months post randomisation
Measurement of quality of life using EQ-5D-5L score | 6 months post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew King, Principal Investigator — University of Manchester
Locations (17):
- United Kingdom (17):
  - Derriford Hospital, Plymouth, Devon
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - University Hospital of Wales, Cardiff, Wales
  - Leeds General Infirmary, Leeds, Yorkshire
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, Bristol
  - Addenbrookes Hospital, Cambridge
  - The Walton Centre, Liverpool
  - Royal London Hospital, London
  - St George's Hospital, London
  - Charing Cross Hospital, London
  - National Hospital for Neurology and Neurosurgery, Queen Square, London
  - Northern Care Alliance NHS Foundation Trust, Manchester
  - Queens Medical Centre, Nottingham
  - Royal Preston Hospital, Preston
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent